CLINICAL TRIAL: NCT05591300
Title: Microparticles Blood Level in Acute Carbon Monoxide Poisoning
Acronym: COMPs
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Collaborators: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Responsible Party: Principal Investigator, Rosanna Vaschetto, MD, PhD, Professor, Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: AOCarita1
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Carbon Monoxide Poisoning
Keywords: Carbon monoxide intoxication; Microparticles; Microvesicles; Carbon monoxide poisoning; CO; Delayed neurological syndrome; Hyperbaric Oxygen
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 45 Days
Biospecimen Retention: Samples Without DNA — 3 ml blood in sodium citrate before and after hyperbaric treatment will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with acute CO poisoning needing a hyperbaric oxygen treatment
  Interventions: Diagnostic Test: Microparticles research
- Healthy controls: Healthy controls i.e., healthy phisicians than will enter the hyperbaric oxygen therapy chamber to assist the patients
  Interventions: Diagnostic Test: Microparticles research

INTERVENTIONS:
Diagnostic Test: Microparticles research — The absolute count of the total circulating microparticles will be carried out on the patients' plasma using the NanoSight NS300 instrument (Alphatest). Furthermore, the circulating microparticles will be stained with a combination of three monoclonal antibodies (Becton and Dickinson, NJ,USA) to detect microparticles released by the most abundant cell populations in the blood: leukocyte-derived microparticles (CD45+), endothelial-derived microparticles (CD31+), and PLT-derived microparticles (CD31+ CD41a+).

SUMMARY:
The goal of this pilot, clinical, experimental, biological and prospective study with uso of biological material (venous blood sampling), in patient with acute carbon monoxide (CO) intoxication and in a group of healthy non-intoxicated subject (group of control) is the research of a possible increase of circulating microparticles level in human blood with an acute carbon monoxide intoxication.

The main question to answer is:

Is there an increase of circulating microparticles levels in subjects with acute carbon monoxide poisoning? Two blood samples will be withdrawn from patients with acute carbon monoxide poisoning, one before and one after hyperbaric oxygen treatment.

Researchers will compare a group of healthy volunteers to see if there is a different in circulating microparticles blood level compared to patients with intoxication.

DETAILED DESCRIPTION:
Few agents cause suffering like carbon monoxide (CO) in the humans. The CO pathophysiological mechanism extends beyond the hypoxic stress given by the COHb, and current knowledge cannot explain all of the lesions.

CO toxicity includes hypoxic and oxidative stress and implies long-term neurological morbidity. Patients exposed for a short time even to low concentrations of CO may show activation of intravascular neutrophils and increases in circulating inflammatory proteins.

The treatment of CO poisoning is administer normobaric or hyperbaric oxygen. One of the possible complications of CO poisoning is the delayed neurological syndrome.

Microvesicles are microparticles released by all eukaryotic cells and are involved in the intracellular communication, in physiological and pathological conditions.

In the human blood microparticles are present after exposure to tobacco smoke and air pollution.

Mouse model study proved the increased number of circulating microparticles in mice subjected to CO intoxication. Our study group hypothesized a possible increase of circulating microparticles in patient with CO poisoning compared to a population of healthy controls. Secondary objectives will be to assess the relationship between severity of intoxication and circulating microparticles level; risk fatcors for development of delayed neurological syndrome will be investigated. Finally, the types of microparticles involved in CO poisoning will be characterized.

The study population consists by all patients who need a hyperbaric treatment due to an acute CO poisoning in the region afferent to Nursing House Habilita "I Cedri", located in Fara Novarese; for every two patient a healty control will be identified.

When the patient will arrived in hyperbaric room, before the treatment (T0-time zero) a blood sample in sodium citrate will be taken, at the end of the treatment (T1-time one) another blood sample will be taken. The blood samples will then be sent to the laboratory of the Novara Hospital for the processing.

It will be administered a questionnaire for the mental status evaluation (Pfeiffer's Test) in T0 and 45 days after intoxication (T2-time two) by phone to assess the onset of delayed neurological syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Acute carbon monoxide poisoning
* Need for treatment with hyperbaric oxygen

Exclusion Criteria:

* Patient reject to consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with CO poisoning that need hyperbaric oxygen treatment and afferent to the Hyperbaric center of the Nursing Home Habilita "I Cedri" located in Fara Novarese (NO). For every two intoxicated patients it will be necessary identify a healthy volunteer (matching 2:1) comparable with the patient intoxicated by sex, age (+/- 5 years), cigarette smoke.
Sampling Method: Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Microparticles research | 2 years
  Quantify the number and the type of circulating microparticles in subjects after carbon monoxide poisoning.

SECONDARY OUTCOMES:
Relationship between poisoning severity and circulating microparticles levels | 45 days
  Evaluate the possible relationship between carbon monoxide poisoning severity measured as COHb levels and circulating microparticles levels before and after hyperbaric oxygen treatment.
Risk factors of delayed neurological syndrome development | 45 days
  Research of risk factors of delayed neurological syndrome development and follow up with test of Pfeiffer.
Proteomic and transcriptomic analysis | 2 years
  Researche the type of microparticles with proteomic and transcriptomic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna Vaschetto, MD, PhD, Principal Investigator — University of Eastern Piedmont
Locations (1):
- AOU Maggiore della Carità, Novara, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data properties will be maintained by the center involved in the study. Pseudonymized data will not be transferred in other countries outside European Union. Principal investigator will considered data shearing after reasonable request.